CLINICAL TRIAL: NCT01003353
Title: Maximal Strength Training for Chronic Phase Stroke Patients
Brief Title: Strength Training for Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009/1241
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Stroke
Keywords: Stroke; Strength training; exercise therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Maximal strength training — Training will be carried out 3 times a week for 8 weeks. Each session will include a warm up, strength training and warm down. The total time will be approximately 1 hour. The training will consist 2 exercises (leg press and plantarflexion). Participants will train each leg individually with 4 sets of 4 repetitions at 90% of the 1 repetition maximum.

SUMMARY:
The study aims to investigate the effects of strength training on maximal strength, walking ability and neural function in chronic stroke patients. The strength training intervention in this study is different to all previous interventions for stroke patients.

Maximal Strength Training (MST) involves weights of up to 90% of the participants 1 repetition maximum and has a focus on the explosive development of force. This study will use these principles for unilateral leg press and plantarflexion exercises. Only 2 previous studies have investigated high intensity strength training for stroke patients and they used intensities of 80% 1RM. Previous MST interventions have shown large increases in strength, rate of force development and this has transferred to improved walking economy.

The investigators predict that MST will give large increases in strength, improved rate of force development (RFD) and walking economy. The investigators expect that better neural function will account for the improvements. This study could provide evidence for the adoption of a completely different method of strength rehabilitation for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Under 67 years old
* Suffered from a stroke at least 6 months previously
* Living in the Trondheim area such that travel costs can be covered by 1500 NOK
* Must be able to walk, although use of aids is permitted

Exclusion Criteria:

* Participants must not have cognitive, visuospatial or comprehension deficits to magnitude such that it interferes with the ability to perform testing and training
* Participants must be medically unstable (e.g. uncontrollably high blood pressure (140/90), arrythmia, other heart instabilities or other known comorbid diseases)
* Participants must not be known to be pregnant

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Unilateral 1 repetition maximum for leg press and plantarflexion | November 2009-March 2010

SECONDARY OUTCOMES:
Rate of force development in unilateral leg press and plantarflexion | November 2009 - March 2010
Maximal oxygen uptake and walking economy | November 2009 - March 2010
Timed Up and Go Test | November 2009 - March 2010
4 Step Balance Test | November 2009 - March 2010
V-Wave (using sEMG equipment) of soleus during static plantarflexion | November 2009 - March 2010
Blood lipid profile | November 2009 - March 2010
6 Minute Walk Test | November 2009 - March 2010
Jump Height of a countermovement jump | November 2009 - March 2010
SF-36 Quality of life questionnaire, Norwegian version | November 2009 - March 2010

CONTACTS AND LOCATIONS:
Overall Officials: Tom Tørhaug, MD, Principal Investigator — St.Olav's University hospital; Jan Hoff, PhD, Study Chair — National Taiwan Normal University; Jan Helgerud, Principal Investigator — National Taiwan Normal University; Tor Ivar Gjellesvik, Principal Investigator — National Taiwan Normal University; Marius Fimland, Principal Investigator — National Taiwan Normal University; Per Marius R Moen, Principal Investigator — National Taiwan Normal University; Tessa Hill, Principal Investigator — National Taiwan Normal University
Locations (1):
- Avdeling for ervervede hjerneskader, Klinikk for fysikalsk medisin og rehabilitering, St Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Result] Hill TR, Gjellesvik TI, Moen PM, Torhaug T, Fimland MS, Helgerud J, Hoff J. Maximal strength training enhances strength and functional performance in chronic stroke survivors. Am J Phys Med Rehabil. 2012 May;91(5):393-400. doi: 10.1097/PHM.0b013e31824ad5b8. PMID 22357133